CLINICAL TRIAL: NCT04595526
Title: Optimal Collection of Specimens of the Lower Respiratory Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHS-ED-08-2020
Record Dates: First submitted 2020-08-31; First posted 2020-10-20 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tracheal suction (Active Comparator): Uses the local standard procedure of tracheal suction to obtain secretions from the lower respiratory tract
  Interventions: Procedure: Tracheal suction
- Forced expiratory technique and induced sputum (Experimental): This procedure is without suction. The patient's attempts to deliver a sputum sample after forced exhalation and coughing technique. Regardless of the result the patient then receives hypertonic saline by an inhalation mask to induce the sputum. If the patient cannot deliver a sample, tracheal suction will be performed in order to obtain a specimen for the analyses.
  Interventions: Procedure: Forced expiratory technique and induced sputum

INTERVENTIONS:
Procedure: Forced expiratory technique and induced sputum — The intervention is based on the patient's own attempt to deliver a sputum sample after instructions of proper huff forced exhalation and coughing technique. After an attempt to deliver a sputum sample the patient will receive a 0,9% isotonic saline by an inhalation mask to induce the sputum, thereafter the patient will again make an effort to expectorate a sputum sample repeating the forced expiratory technique.
  Arms: Forced expiratory technique and induced sputum
Procedure: Tracheal suction — Tracheal suction is often used on intubated patients at the intensive care unit to collect sputum, and this method has become the standard procedure at several emergency departments.
  Arms: Tracheal suction

SUMMARY:
Respiratory tract infection is a serious condition causing 3 million deaths worldwide every year. Approximately 20-40% of patients with community-acquired pneumonia are hospitalised. Treatment of pneumonia should be initiated as quickly as possible and therefore an early and precise diagnostic is extremely important. Imprecise or delayed diagnosis often results in overconsumption of broad-spectrum antibiotics that contribute to the development of antibiotic resistance. Unspecific symptoms, unsure diagnosis methods and a wait time of up to several days for results challenge a quick and effective diagnosis and treatment of pneumonia. Microbiological analysis of sputum samples is used to identify pathogens causative to pneumonia. However, obtaining specimens of good quality is challenging and affects the sensitivity and specificity of the results. Therefore, the identification of the optimal sputum collecting method is needed to ensure an improved identification process of the pathogen causing pneumonia.

The purpose of this study is to determine the most optimal method for obtaining good quality sputum samples when comparing tracheal suction to methods without suction. A more accurate diagnosis will lead to more appropriate antibiotic consumption and will reduce the general development of antibiotic resistance.

DETAILED DESCRIPTION:
Multi-resistant bacteria (MRB) are associated with high antibiotic consumption and designated by WHO as one of the major threats to the world. In Denmark, the incidence of MRB is generally increasing, and every 20th patient admitted to Danish Emergency Department (ED), is infected with resistant bacteria. Respiratory tract infection is a serious condition, with 3 million death worldwide every year, and about 20-40% of the patients with community-acquired pneumonia need hospitalization. Data from the ED at Hospital Sønderjylland shows that 6% of the patients are registered with a respiratory tract infection, including pneumonia. Treatment of pneumonia should be initiated within a few hours, therefore early and precise diagnostic is extremely important. An imprecise or delayed diagnostic will often result in overconsumption of broad-spectrum antibiotics, contributing to an increase in the development of MRB threatening future treatments possibilities. Currently, pneumonia diagnosis is based on clinical symptoms such as cough, expectoration, chest pain, fever or breathlessness, combined with an x-ray of the lungs, relevant blood tests and microbiological analyses of sputum samples. However, X-ray is an imprecise diagnostic tool, and sputum test responses are first available after 2 days. Thus, the diagnostic is challenged by unspecific symptoms, unsure diagnostic methods and prolonged waiting time for results of up to several days. Sputum can be cultivated to determine the bacterial agent. However, the sputum samples are often of poor quality and many patients cannot deliver a sample. A recently published Danish study shows, that only half of the patients at the ED have sputum samples collected for culturing and none of them had their antibiotic treatment adjusted based on the microbiological results of the sputum. Despite, the use of different microbiological analysis methods to detect bacteria or virus causative of pneumonia, common to the methods is that a representative specimen from the lower respiratory tract is crucial for optimal sensitivity and specificity. Despite technological advances in molecular diagnostics, identifying the etiology of pneumonia remains a challenge. Consequently, identification of optimal sputum collecting method and investigation of an alternative sputum analyses assessment is needed to improve specimens' suitability to identify the etiology of pneumonia.

Clinical experience indicates that an inhalation mask with saline solution can induce a successful sputum sampling. Tracheal suction is often used on intubated patients in the intensive care unit to collect sputum, and this method has become the standard procedure at several ED. A comparison of the two methods has not been investigated in an ED context nor has the quality of the collected sputum samples and relevance for clinical practice been explored.

Ensuring the optimal sputum collection is of particular relevance during the COVID-19 pandemic. An optimal sputum collection is important to be able to determine if the pneumonia is caused by SARS-CoV-2 or a bacterium - especially in situations where the swab from throat or pharynx presents a negative result, as the method is not sensitive enough to rule out COVID-19 in patients with pneumonia. Accordingly, the Health Board in Denmark recommends tracheal suction of patients admitted with suspected COVID-19 in case of symptoms of the lower respiratory tract, and only in cases the symptoms originates from the upper airways a swab can be performed

1.1 Hypothesis and purpose The hypotheses is that methods without suction (forced expiratory technique and induced sputum) are just as effective as tracheal suction for obtaining a representative specimen from the lower respiratory tract..

The purpose of this study is to determine the most optimal method for obtaining high-quality sputum samples.

Following research questions will be explored:

1. What is the difference between the conventional sampling by tracheal suction comparing to sampling using forced expiratory or induced sputum techniques in relation to the suitability of collected specimens from the lower respiratory tract
2. Identification of possible adverse events during sputum collection
3. How do patients experience the two sputum sample collecting procedures?

Collection of sputum and adverse events After consent, the patient will be randomized in two groups with 1:1 allocation using permuting blocks. The software tool 'Randomized' offered by Open Patient data Explorative Network (OPEN) will be used.

ORGANIZATION The project is anchored in the Research unit of Emergency Medicine, the ED of Hospital Sønderjylland and the Department of Regional Health Research, University of Southern Denmark. The project is a research collaboration between clinicians and researchers in the field of emergency medicine and microbiology at Hospital Sønderjylland (SHS) and Odense University Hospital (OUH).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with suspected lower respiratory tract infection
* Patients > 18 years old
* One of the following symptoms: dyspnea, cough, expectoration, fever and chest tightness

Exclusion Criteria:

* Patients transferred directly to ICU
* If the attending physician considers emergency treatment is needed
* Patients receiving prednisolone treatment of 20mg/day or more over the last 2 weeks
* Patient which consent cannot be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Quality of specimen from the lower respiratory tract | From collection to culture results - up to 5 days
  Unsuitable (bad quality) measured by microscopy - > 10 squamous epithelial cells per low power field of view (x10). Suitable (good quality) measured by microscopy - Samples with < 10 squamous epithelial cells per low power field of view

SECONDARY OUTCOMES:
Patient clinical symptoms | Patients are followed before intervention and 10 minutes after intervention
  The patients are asked about 4 specific symptoms (Cough, Expectoration, Chest pain and Dyspnea). The clinical symptoms are measured as following: yes/no/yes worse than usual. Ten minutes after the intervention they will be asked the same questions with yes/no/worse than before the intervention.
Respiratory rate | Measured twice: Baseline ( at admission) and follow up (10 minutes after intervention)
  This will be counted by the health professional attending the patient and is the number of breaths per minute in rest. It is assessed by counting the number of times the patients chest rises in a half minute multiplied by 2.
Oxygen saturation | Measured twice: Baseline ( at admission) and follow up (10 minutes after intervention)
  This is measured using a pulse oximetry device - a non-invasive method to measure arterial oxygen saturation level in percentages
Patient well-being and experience of procedure | Measured twice: Baseline ( at admission) and follow up (10 minutes after intervention)
  Measured using the Borg Categorical rate 10 scale and a single likert-scale question - 'How does the patient experience the procedure' (only measured after the intervention).
Occurrence of side effects | Registered up to 1 hour after intervention
  Project assistants will register any side effects such as bleeding from the airways and bronchospasm.
Short term mortality | Registered within 7 days from hospital admission
  Death within 7 days from hospital admission
Number of patients readmitted to hospital | Registered within 1 month after readmission
  30 days readmission after current hospitalization
Patient experience of sputum collection | Measured 5 minutes after procedure
  This outcome will be measured once after an attempt at sputum collection. A five-point Likert scale ranging from "very bad, bad, neither bad nor good, good, very good" will be used to report how the patient experienced the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, MD PhD, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Overend TJ, Anderson CM, Brooks D, Cicutto L, Keim M, McAuslan D, Nonoyama M. Updating the evidence-base for suctioning adult patients: a systematic review. Can Respir J. 2009 May-Jun;16(3):e6-17. doi: 10.1155/2009/872921. PMID 19557211
- [Background] Skjot-Arkil H, Mogensen CB, Lassen AT, Johansen IS, Chen M, Petersen P, Andersen KV, Ellermann-Eriksen S, Moller JM, Ludwig M, Fuglsang-Damgaard D, Nielsen FE, Petersen DB, Jensen US, Rosenvinge FS. Carrier prevalence and risk factors for colonisation of multiresistant bacteria in Danish emergency departments: a cross-sectional survey. BMJ Open. 2019 Jun 27;9(6):e029000. doi: 10.1136/bmjopen-2019-029000. PMID 31253624
- [Background] Meehan TP, Fine MJ, Krumholz HM, Scinto JD, Galusha DH, Mockalis JT, Weber GF, Petrillo MK, Houck PM, Fine JM. Quality of care, process, and outcomes in elderly patients with pneumonia. JAMA. 1997 Dec 17;278(23):2080-4. PMID 9403422
- [Background] Karakioulaki M, Stolz D. Biomarkers and clinical scoring systems in community-acquired pneumonia. Ann Thorac Med. 2019 Jul-Sep;14(3):165-172. doi: 10.4103/atm.ATM_305_18. PMID 31333765
- [Background] Savvateeva EN, Rubina AY, Gryadunov DA. Biomarkers of Community-Acquired Pneumonia: A Key to Disease Diagnosis and Management. Biomed Res Int. 2019 Apr 30;2019:1701276. doi: 10.1155/2019/1701276. eCollection 2019. PMID 31183362
- [Background] Saukkoriipi A, Palmu AA, Jokinen J. Culture of all sputum samples irrespective of quality adds value to the diagnosis of pneumococcal community-acquired pneumonia in the elderly. Eur J Clin Microbiol Infect Dis. 2019 Jul;38(7):1249-1254. doi: 10.1007/s10096-019-03536-9. Epub 2019 Apr 4. PMID 30949897
- [Background] Miyashita N, Shimizu H, Ouchi K, Kawasaki K, Kawai Y, Obase Y, Kobashi Y, Oka M. Assessment of the usefulness of sputum Gram stain and culture for diagnosis of community-acquired pneumonia requiring hospitalization. Med Sci Monit. 2008 Apr;14(4):CR171-6. PMID 18376343
- [Background] Murdoch DR. How best to determine causative pathogens of pneumonia. Pneumonia (Nathan). 2016 Apr 12;8:1. doi: 10.1186/s41479-016-0004-z. eCollection 2016. PMID 28702281
- [Background] Herrero-Cortina B, Alcaraz V, Vilaro J, Torres A, Polverino E. Impact of Hypertonic Saline Solutions on Sputum Expectoration and Their Safety Profile in Patients with Bronchiectasis: A Randomized Crossover Trial. J Aerosol Med Pulm Drug Deliv. 2018 Oct;31(5):281-289. doi: 10.1089/jamp.2017.1443. Epub 2018 Jun 7. PMID 29878856
- [Derived] Cartuliares MB, Skjot-Arkil H, Rosenvinge FS, Mogensen CB, Skovsted TA, Pedersen AK. Effectiveness of expiratory technique and induced sputum in obtaining good quality sputum from patients acutely hospitalized with suspected lower respiratory tract infection: a statistical analysis plan for a randomized controlled trial. Trials. 2021 Oct 2;22(1):675. doi: 10.1186/s13063-021-05639-1. PMID 34600559